CLINICAL TRIAL: NCT03472053
Title: A Randomized Study of the Safety and Efficacy of BIO-11006 in Treatment of Advanced Non-Small Cell Lung Cancer in Patients Who Are Not Candidates for Curative Surgery and/or Radiation and Who Are Receiving Pemetrexed and Carboplatin
Brief Title: A Study of BIO-11006 in the Treatment of Advanced Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioMarck Pharmaceuticals, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIO-NSCLC-001
Record Dates: First submitted 2018-03-01; First posted 2018-03-21 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Non Small Cell Lung Cancer Stage IIIB
Keywords: Lung cancer; non small cell; metastasis
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Neoplasm Metastasis | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Patients will be randomized in 1:1 ratio to either BIO-11006 plus Standard of Care (intervention) or Standard of Care (Pemetrexed plus Carboplatin) (intervention).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BIO-11006 plus standard of care (Experimental): Aerosolized BIO-11006 (125mg BID) plus standard of care (Pemetrexed plus Carboplatin) is administered for three months.
  Interventions: Drug: BIO-11006 plus standard of care
- Standard of Care (Experimental): Pemetrexed (500 mg/meter square) and Carboplatin (AUC6, Calvert's Formula) is administered every three weeks for three months.
  Interventions: Drug: Standard of Care

INTERVENTIONS:
Drug: BIO-11006 plus standard of care — BIO-11006 is administered 125mg BID plus standard of care.
  Other Names: Active drug plus standard of care
  Arms: BIO-11006 plus standard of care
Drug: Standard of Care — Pemetrexed (500 mg/meter square) and Carboplatin (AUC6, Calvert's formula) are administered every three weeks for three months.
  Other Names: Active comparator
  Arms: Standard of Care

SUMMARY:
This Phase 2 is a randomized study in advanced Non-Small Cell lung cancer patients to evaluate safety and efficacy of aerosolized BIO-11006 in conjunction with chemotherapy.

DETAILED DESCRIPTION:
This randomized, open label, multicenter Phase 2 study is to evaluate safety and efficacy of BIO-11006 in Stage IIIB Non Small Cell Lung cancer (NSCLC) patients who are not candidates for curative surgery, radiation, or immunotherapy and who are also receiving Pemetrexed and Carboplatin as standard of care (SOC). This study will be conducted at ten clinical centers in India under an IND from US-FDA and an IND from Indian FDA.

This is a parallel 2- Arm study in which a total of 60 patients will be randomized. One Arm of 30 subjects will receive aerosolized 125mg BIO-11006 BID using Pari eFlow nebulizer in conjunction with SOC chemotherapy (Pemetrexed plus Carboplatin). A second Arm of 30 subjects will receive only SOC chemotherapy (Pemetrexed plus Carboplatin). The treatment period will be three months and nine months survival follow up period (every three months).

Primary efficacy endpoint will be Progression-free survival (PFS) in patients who receive BIO-11006 plus SOC compared to those who receive SOC alone. The secondary efficacy endpoints will include: a. Response rate at three months (4 cycles) per RECIST V1.1; (b) overall survival; and (c) patient body weight maintenance.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are physically able to self administer drug by nebulizer;
2. Measurable disease per RECIST Version 1.1;
3. Female patients of child bearing age must have a negative pregnancy test;
4. ECOG 0-2;
5. Written informed consent;

Exclusion Criteria:

1. Candidates for curative surgery and/or radiation therapy;
2. Baseline ANC<2000 cells/mm cube; platelet count <100,000 cells/mm cube
3. Creatinine clearance <45 mL/min;
4. Billirubin >2 x the upper limit of normal
5. Known history of HIV, hepatitis B, hepatitis C or tuberculosis;
6. Current pneumonia or idiopathic pulmonary fibrosis;
7. Hypersensitivity to test drug, pemetrexed, or carboplatin.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | 12 months
  Survival period of patients in both arms of the study is measured in absence of tumor progression.

SECONDARY OUTCOMES:
Maintenance of body weight | 3 and12 months
  Patient's body weight in kilograms measured at three month and at 12 month to assess possible disease related cachexia.
Treatment emergent adverse effects | 3 months
  Treatment-emergent adverse events including headache, bronchitis, dyspnea, cough, pyrexia, chest discomfort and liver function will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Devesh Verma, PhD, Study Director — Cliantha Research India
Locations (11):
- India (11):
  - Unique Hospital and Research Institute, Surat, Gujarat
  - Aadhar Health Institute, Hisar, Haryana
  - Chirayu Cancer Hospital, Bhopal, Madhya Pradesh
  - Tata Memorial Hospital, Mumbai, Maharashtra
  - Navsanjeevani Hospital, Nashik, Maharashtra
  - HCG Manavata Cancer Center, Nashik, Maharashtra
  - Deenanath Mangeshkar Hospital & Research Center, Pune, Maharashtra
  - Vardhman Mahavir Medical College & Hospital, New Delhi, National Capital Territory of Delhi
  - Sparsh Hospitals and Critical Care, Bhubaneswar, Odisa
  - SMS Medical College & Hospital, Jaipur, Rajasthan
  - Nehru Hospital & Post Graduate Institute of Medical Education, Chandigarh

IPD SHARING:
Plan to Share IPD: Undecided